CLINICAL TRIAL: NCT00710060
Title: NIMH Collaborative HIV/STD Prevention Trial
Brief Title: Effectiveness of a Community-level HIV/STD Prevention Intervention in Promoting Safer Sexual Behaviors in High-risk Populations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Willo Pequegnat, PhD/Principal Investigator, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U10MH061537 (NIH); U10MH061537 (NIH); U10MH061499 (NIH); U10MH061513 (NIH); U10MH061536 (NIH); U10MH061543 (NIH); U10MH061544 (NIH); DAHBR 9A-ASGT
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2008-07

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: HIV; Popular Opinion Leader; POL; Behavioral Intervention; STD; STI; Community; Prevention; International; Global
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participating communities will receive the Community Popular Opinion Leader intervention and HIV/STD educational materials.
  Interventions: Behavioral: Community Popular Opinion Leader (C-POL); Behavioral: HIV/STD educational materials
- 2 (Active Comparator): Participating communities will receive HIV/STD educational materials only.
  Interventions: Behavioral: HIV/STD educational materials

INTERVENTIONS:
Behavioral: Community Popular Opinion Leader (C-POL) — The C-POL intervention will teach identified opinion leaders to share personalized HIV prevention messages in conversations with peers in an effort to change community norms. Opinion leaders will be taught skills for sharing HIV risk-reduction messages during four to five weekly training sessions. At least 15% of the community population will be trained as opinion leaders. After the initial training, opinion leaders will attend six to nine booster sessions over the next 2 years to reinforce and support continued conversation efforts.
  Other Names: Popular Opinion Leader (POL); Diffusion of Innovations
  Arms: 1
Behavioral: HIV/STD educational materials — Communities will receive HIV/STD educational materials and treatment referral information to distribute to community members.

SUMMARY:
This study will evaluate the effectiveness of a community-level HIV prevention program in promoting safer sexual behaviors and reducing the transmission of HIV/sexually transmitted diseases among at-risk populations in China, India, Peru, Russia, and Zimbabwe.

DETAILED DESCRIPTION:
The HIV/AIDS epidemic remains largely out of control in many areas of the world, with an estimated 2.5 million new HIV infections worldwide in 2007. Developing countries with few economic resources and world regions undergoing difficult social transitions have been particularly impacted by large increases in HIV and sexually transmitted disease (STD) infections. To date, effective individual prevention approaches have not been rapid enough to avert the epidemic in these areas and may be too resource intensive to maintain. Behavioral HIV prevention interventions on the community level seek to reduce the prevalence of high-risk sexual behaviors by reaching large numbers of vulnerable people in a cost-effective and feasible manner, even in areas with limited resources. The Community Popular Opinion Leader (C-POL) program is an HIV prevention intervention that recruits and trains trusted opinion leaders in the community to promote safe sex behaviors through risk-reduction conversations with peers. Implementing the C-POL program in world regions facing significant HIV/AIDS epidemics may be the most effective means of encouraging behavior change among members of at-risk populations and strengthening social norms to maintain these changes. This study will evaluate the effectiveness of the C-POL program in promoting safer sexual behaviors and reducing the transmission of HIV/STDs among at-risk populations in China, India, Peru, Russia, and Zimbabwe.

Participation in this study will last 2 years. Initially, an ethnographic study will be conducted to determine the HIV/STD knowledge, attitudes, and behaviors among the population living in the target communities. Information collected via observation, focus groups, and interviews will be used to determine the social risk groups operating within the community and to identify and recruit the opinion leaders who are influential in these groups. Also, an epidemiological study will be conducted to collect information on sexual behaviors and HIV/STD rates.

A cohort of members from participating communities will first undergo baseline assessments that will include a survey about general health and knowledge of HIV/STDs and a biological sampling for HIV/STD testing. Participating communities will then be assigned randomly to receive the C-POL intervention and HIV/STD educational materials or HIV/STD educational materials alone. In communities receiving the C-POL intervention, the previously recruited opinion leaders will be taught skills for sharing HIV risk-reduction messages in daily conversation with peers. This training will occur over four to five weekly sessions. At least 15% of the community population will be trained as opinion leaders. After the initial training, opinion leaders will attend six to nine booster sessions over the next 2 years to reinforce and support continued conversation efforts. Communities assigned to receive the HIV/STD educational materials will receive informational materials on HIV/STDs to provide to community members and will provide treatment or treatment referral for people with nonviral STDs.

All participants in the baseline cohort will be asked to repeat the baseline testing 1 and 2 years later. Participants who are not able to visit a clinic for testing will be contacted by phone to complete the baseline survey. After the 2-year assessments, the C-POL intervention will be conducted in the communities that received educational materials only.

ELIGIBILITY:
Inclusion Criteria:

* Either lives, works, or socializes in the selected venues
* Plans to remain in the venue for at least 1 year after study entry

Exclusion Criteria:

* Permanent disability that hinders participation (e.g. deaf, mental retardation)
* Reports no sex in the 6 months before study entry (China, Peru)
* No STDs present at study entry (China)
* Enrolled in final year of school at time of recruitment (Russia)
* Has lived in venue for less than 2 years (Zimbabwe)
* Lives in venue for less than 9 months out of a year (Zimbabwe)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18147 (Actual)
Dates: Start 2002-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected sexual acts with nonspousal partners | Measured at baseline and Years 1 and 2
Overall observed incidence of sexually transmitted diseases (STDs) (e.g., chlamydia, gonorrhea, syphilis, trichomonas, HIV, or herpes simplex virus-2), as detected by biological specimens | Measured at baseline and Years 1 and 2

SECONDARY OUTCOMES:
Increased exposure to HIV prevention messages, more STD treatment seeking, lower stigma regarding HIV and STDs, and lower substance abuse associated with sexual behavior in intervention group as compared to control group | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Carlos F. Caceres, PhD, Principal Investigator — Cayetano Heredia University, Lima, Peru; David D. Celentano, ScD, Principal Investigator — The Johns Hopkins University, Baltimore, Maryland (India); Thomas J. Coates, PhD, Principal Investigator — University of California at Los Angeles, Los Angeles, California (Peru); Tyler D. Hartwell, PhD, Principal Investigator — RTI International, Research Triangle Park, North Carolina (DCC); Danuta Kasprzyk, PhD, Principal Investigator — Battelle Center for Public Health Research and Evaluation, Seattle, Washington (Zimbabwe); Jeffrey A. Kelly, PhD, Principal Investigator — Medical College of Wisconsin, Milwaukee, Wisconsin (Russia); Andrei P. Kozlov, PhD, Principal Investigator — Biomedical Center, St. Petersburg State University, St. Petersburg, Russia; Willo Pequegnat, PhD, Principal Investigator — National Institute of Mental Health, Bethesda, Maryland; Mary Jane Rotheram-Borus, PhD, Principal Investigator — University of California at Los Angeles, Los Angeles, California (China); Suniti Solomon, MD, Principal Investigator — YRG Centre for AIDS Research and Education, Chennai, India; Godfrey B. Woelk, PhD, Principal Investigator — University of Zimbabwe Medical School, Harare, Zimbabwe; Zunyou Wu, MD, PhD, Principal Investigator — Chinese Center for Disease Control and Prevention, Beijing, P.R. China
Locations (5):
- Fujian Institute of Health Education, Fuzhou, China
- YRG Centre for AIDS Research and Education (YRGCARE), Chennai, India
- Universidad Peruana Cayetano Heredia, Lima, Peru
- Biomedical Center, Saint Petersburg, Russia
- Zimbabwe Community Health Intervention Research (ZiCHIRe) - University of Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Methodological overview of a five-country community-level HIV/sexually transmitted disease prevention trial. AIDS. 2007 Apr;21 Suppl 2:S3-18. doi: 10.1097/01.aids.0000266453.18644.27. PMID 17413262
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Selection of populations represented in the NIMH Collaborative HIV/STD Prevention Trial. AIDS. 2007 Apr;21 Suppl 2:S19-28. doi: 10.1097/01.aids.0000266454.26268.90. PMID 17413260
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Challenges and processes of selecting outcome measures for the NIMH Collaborative HIV/STD Prevention Trial. AIDS. 2007 Apr;21 Suppl 2:S29-36. doi: 10.1097/01.aids.0000266455.03397.08. PMID 17413261
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Design and integration of ethnography within an international behavior change HIV/sexually transmitted disease prevention trial. AIDS. 2007 Apr;21 Suppl 2(Suppl 2):S37-48. doi: 10.1097/01.aids.0000266456.03397.d3. PMID 17413263
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. The feasibility of audio computer-assisted self-interviewing in international settings. AIDS. 2007 Apr;21 Suppl 2(Suppl 2):S49-58. doi: 10.1097/01.aids.0000266457.11020.f0. PMID 17413264
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. The community popular opinion leader HIV prevention programme: conceptual basis and intervention procedures. AIDS. 2007 Apr;21 Suppl 2:S59-68. doi: 10.1097/01.aids.0000266458.49138.fa. PMID 17413265
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Ethical issues in the NIMH Collaborative HIV/STD Prevention Trial. AIDS. 2007 Apr;21 Suppl 2(Suppl 2):S69-80. doi: 10.1097/01.aids.0000266459.49138.b3. PMID 17413266
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Sexually transmitted disease and HIV prevalence and risk factors in concentrated and generalized HIV epidemic settings. AIDS. 2007 Apr;21 Suppl 2:S81-90. doi: 10.1097/01.aids.0000266460.56762.84. PMID 17413267
- [Background] NIMH Collaborative HIV/STD Prevention Trial Group. Formative study conducted in five countries to adapt the community popular opinion leader intervention. AIDS. 2007 Apr;21 Suppl 2:S91-8. doi: 10.1097/01.aids.0000266461.33891.d0. PMID 17413268
- [Background] NIMH Collaborative HIV/STD Prevention Trial. Role of the data safety and monitoring board in an international trial. AIDS. 2007 Apr;21 Suppl 2(Suppl 2):S99-102. doi: 10.1097/01.aids.0000266462.33891.0b. PMID 17413269
- [Derived] Rotheram-Borus MJ, Wu Z, Liang LJ, Li L, Detels R, Guan J, Yin Y, Swendeman D; NIMH Collaborative HIV/STD Prevention Trial Group. Reductions in sexually transmitted infections associated with popular opinion leaders in China in a randomised controlled trial. Sex Transm Infect. 2011 Jun;87(4):337-43. doi: 10.1136/sti.2010.046243. Epub 2011 Jan 29. PMID 21278400
- See also: Click here for more information on this study at the NIMH Collaborative HIV/STD Prevention Trial Web site — http://www.rti.org/u10